CLINICAL TRIAL: NCT00544414
Title: Multimodality Management of Head and Neck Cancer: A Phase II Trial of Induction Chemotherapy, Organ Preservation Surgery, and Concurrent Chemoradiotherapy
Brief Title: Chemotherapy Followed by Surgery, Chemotherapy, and Radiation Therapy in Treating Patients With Locally Advanced Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98147; P30CA033572 (NIH); CHNMC-98147; CDR0000566884 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel; Fluorouracil; Gemcitabine; Leucovorin; Gene Expression Profiling; Chemotherapy, Adjuvant; Biopsy; Neoadjuvant Therapy; Radiotherapy

ARMS (1):
- Treatment (Experimental): Patients receive neoadjuvant induction chemotherapy comprising docetaxel IV over 1 hour on day 1 and cisplatin IV, leucovorin IV, and fluorouracil IV over 24 hours on days 1-4. Induction chemotherapy repeats every 28 days for 3 courses.
  Patients with partial response at the primary site may undergo radical or functional resection of the primary tumor within 3 weeks of completion of neoadjuvant therapy.
  Beginning within 4 weeks of completion of neoadjuvant therapy, patients with persistent disease or complete response after chemotherapy at the primary or neck then undergo radiotherapy 5 days a week for 7 weeks and receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 60 minutes on day 1 of each week of radiotherapy.
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: leucovorin calcium; Genetic: gene expression analysis; Genetic: protein expression analysis; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: biopsy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs such as gemcitabine and cisplatin may make tumor cells more sensitive to radiation therapy. Giving combination chemotherapy before surgery or radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving chemotherapy followed by surgery, chemotherapy, and radiation therapy works in treating patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the complete and overall response rate of neoadjuvant docetaxel, cisplatin, fluorouracil, and leucovorin calcium in previously untreated patients with local regionally advanced head and neck cancer.
* To evaluate the feasibility of a multimodality treatment approach with the goal of reducing long-term sequelae.
* To evaluate prospectively, the impact of neoadjuvant chemotherapy, concurrent chemoradiotherapy, and organ preservation surgery on overall survival, time to progression, and pattern of disease recurrence in these patients.
* To evaluate prospectively, biochemical correlates of response and prognosis, including markers such as thymidylate synthetase, ribonucleotide reductase, and ERCC1 (measured by quantitative PCR), p53 (evaluated by IHC), and HPV status and apoptosis (TUNEL assay).

Secondary

* To evaluate treatment-associated morbidity with the use of a quality of life assessment tool.
* To compare the results of diagnostic salivary cytology with those of histopathology at initial diagnosis as well as follow-up in head and neck cancer patients.
* To evaluate the tolerability of combined chemoradiotherapy using gemcitabine and cisplatin after definitive surgery for squamous cell carcinoma of the head and neck.

OUTLINE: Patients receive neoadjuvant induction chemotherapy comprising docetaxel IV over 1 hour on day 1 and cisplatin IV, leucovorin IV, and fluorouracil IV over 24 hours on days 1-4. Induction chemotherapy repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients with partial response at the primary site may undergo radical or functional resection of the primary tumor within 3 weeks of completion of neoadjuvant therapy.

Beginning within 4 weeks of completion of neoadjuvant therapy, patients with persistent disease or complete response after chemotherapy at the primary or neck then undergo radiotherapy 5 days a week for 7 weeks and receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 60 minutes on day 1 of each week of radiotherapy in the absence of disease progression or unacceptable toxicity.

Patients complete the FACT-H&N quality of life questionnaire at baseline and at completion of neoadjuvant therapy.

Tissue biopsies are collected at baseline, periodically during therapy, at surgery, and after radiotherapy. Tissue is examined for gene and protein expression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck, including any of the following subtypes:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
* Stage III or IV disease

  * Stage II carcinoma of the larynx, hypopharynx, or base of tongue allowed
* Measurable disease
* Resectable disease, defined as tumors that are potentially curable by surgery and radiotherapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 60%
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* Transaminases and alkaline phosphatase meeting 1 of the following criteria:

  * ALT or AST ≤ 2.5 times upper limit of normal (ULN) AND alkaline phosphatase normal
  * Alkaline phosphatase ≤ 4 times ULN AND ALT and AST normal
  * ALT or AST < 1.5 times ULN AND alkaline phosphatase < 2.5 times ULN
* Free of serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior malignancy allowed for purposes of determining disease-free or overall survival except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for 5 years
* No unstable angina, history of congestive heart failure, or acute myocardial infarction within the past 6 months
* No current symptomatic, neurosensory or neuromotor toxicity ≥ grade 2
* No other significant medical or psychiatric condition incompatible with the protocol

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for head and neck cancer

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-06-07 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I. Shibata, MD, Study Chair — City of Hope Comprehensive Cancer Center

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 62 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Hispanic | 6
  White Non-Hispanic | 22
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Complete response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions. Partial response (PR): Greater than or equal 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No new lesions. All measurable and evaluable lesions and sites must be assessed using the same techniques as baseline. Overall Response (OR) = CR + PR.
Time Frame: 30 days after last course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 28

2. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression defined as a 50% increase or an increase of 10 cm^2 (whichever is smaller) in the sum of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or reappearance of any lesion that had disappeared, or appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition. Progression-free survival defined as from first day of treatment until the date of first documented progression or date of death from any cause, whichever came first. If failure has not occurred, failure time is censored at the time of last follow-up.
Time Frame: From date of initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 171 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment
Number analyzed (Participants) | 31
Months | 170.5 [113.3 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 3 years and 9 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 18/31
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 (1)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain - Other (Specify, __) (General disorders) | 1 (2)
Infection with unknown ANC (Infections and infestations) | 2 (3)
Mucositis due to radiation (Injury, poisoning and procedural complications) | 2 (2)
Creatinine (Investigations) | 2 (2)
Leukocytes (total WBC) (Investigations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=31)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1)
Pain due to radiation (General disorders) | 4 (5)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Infections and infestations) | 2 (3)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 31 (100)
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 4 (7)
Transfusion: Platelets (Blood and lymphatic system disorders) | 3 (3)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 7 (8)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 3 (7)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 2 (5)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 24 (50)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 8 (11)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 21 (38)
Diarrhea (Gastrointestinal disorders) | 27 (51)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 4 (4)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 16 (20)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 20 (35)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 23 (75)
Heartburn/dyspepsia (Gastrointestinal disorders) | 15 (22)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Incontinence (Gastrointestinal disorders) | 2 (4)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 29 (66)
Nausea (Gastrointestinal disorders) | 27 (81)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 2 (2)
Salivary gland changes/saliva (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 27 (65)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 8 (14)
Edema (General disorders) | 16 (26)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 30 (81)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 11 (17)
Injection site reaction/extravasation changes (General disorders) | 1 (1)
Irritability (children <3 years of age) (General disorders) | 1 (1)
Pain - Other (Specify, __) (General disorders) | 29 (142)
Rigors/chills (General disorders) | 10 (14)
Infection (Infections and infestations) | 1 (1)
Infection - Other (Specify, __) (Infections and infestations) | 1 (2)
Infection with unknown ANC (Infections and infestations) | 2 (2)
Infection without neutropenia (Infections and infestations) | 1 (1)
Infection, Fungal (COH) (Infections and infestations) | 10 (11)
Infection, Viral (COH) (Infections and infestations) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 (2)
Dysphagia-esophageal related to radiation (Injury, poisoning and procedural complications) | 13 (14)
Mucositis due to radiation (Injury, poisoning and procedural complications) | 18 (18)
Rash: dermatitis associated with radiation (Injury, poisoning and procedural complications) | 18 (18)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 17 (27)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 19 (39)
Alkaline phosphatase (Investigations) | 9 (14)
Bilirubin (hyperbilirubinemia) (Investigations) | 4 (6)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 14 (20)
Creatinine (Investigations) | 17 (32)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 6 (9)
Leukocytes (total WBC) (Investigations) | 29 (63)
Lymphopenia (Investigations) | 24 (47)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 21 (40)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
PTT (Partial Thromboplastin Time) (Investigations) | 3 (3)
Platelets (Investigations) | 20 (39)
Weight gain (Investigations) | 5 (10)
Weight loss (Investigations) | 28 (57)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 28 (64)
Anorexia (Metabolism and nutrition disorders) | 28 (73)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 31 (78)
Dehydration (Metabolism and nutrition disorders) | 23 (42)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 28 (67)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 10 (10)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 27 (56)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 15 (26)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 27 (57)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 29 (66)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 7 (9)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 6 (17)
Dizziness (Nervous system disorders) | 19 (23)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (3)
Neurology - Other (Specify, __) (Nervous system disorders) | 10 (17)
Neuropathy: motor (Nervous system disorders) | 15 (23)
Neuropathy: sensory (Nervous system disorders) | 14 (23)
Pain (Nervous system disorders) | 22 (50)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (3)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 (3)
Syncope (fainting) (Nervous system disorders) | 5 (5)
Taste alteration (dysgeusia) (Nervous system disorders) | 11 (15)
Tremor (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 18 (29)
Mood alteration (Psychiatric disorders) | 23 (62)
Personality/behavioral (Psychiatric disorders) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 4 (6)
Urinary frequency/urgency (Renal and urinary disorders) | 7 (8)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 8 (8)
Urine color change (Renal and urinary disorders) | 1 (1)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 13 (18)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 18 (27)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 18 (31)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 7 (7)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (23)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 9 (12)
Flushing (Vascular disorders) | 8 (10)
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 6 (8)
Hypertension (Vascular disorders) | 6 (9)
Hypotension (Vascular disorders) | 16 (23)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT00544414/Prot_SAP_000.pdf